CLINICAL TRIAL: NCT01006018
Title: DPP-4 Inhibition and Thiazolidinedione for Diabetes Mellitus Prevention (DInT DM Study)
Brief Title: DPP-4 Inhibition and TZD for DM Prevention
Acronym: DInT DM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unanticipated delays due to sterilization/stabilization testing of GLP-1.
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Dr. Mary Rhee, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00015390
Record Dates: First submitted 2009-10-27; First posted 2009-11-02 (Estimated); Results first posted 2013-06-07 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Prediabetic State
Keywords: Prediabetic State
MeSH Terms: conditions — Prediabetic State | interventions — Sitagliptin Phosphate; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sitagliptin + Pioglitazone PLACEBO (Experimental): Sitagliptin (DPP-IV inhibitor) 100 mg daily by mouth
  + pioglitazone PLACEBO daily by mouth
  Interventions: Drug: Sitagliptin + Pioglitazone PLACEBO
- Sitagliptin + Pioglitazone (Experimental): Sitagliptin (DPP-IV inhibitor) 100 mg daily by mouth
  + pioglitazone (TZD) 15 mg daily by mouth
  Interventions: Drug: Sitagliptin + Pioglitazone
- PLACEBO (Placebo Comparator): Sitagliptin (DPP-IV inhibitor) PLACEBO daily by mouth
  + pioglitazone (TZD) PLACEBO daily by mouth
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: Sitagliptin + Pioglitazone PLACEBO — Sitagliptin 100 mg tablet daily + Pioglitazone PLACEBO 15 mg capsule daily
  Other Names: Januvia (sitagliptin); Pioglitazone (Actos)
  Arms: Sitagliptin + Pioglitazone PLACEBO
Drug: Sitagliptin + Pioglitazone — Sitagliptin 100 mg tablet daily + Pioglitazone 15 mg capsule daily
  Other Names: Januvia (sitaglitin); Pioglitazone (Actos)
  Arms: Sitagliptin + Pioglitazone
Drug: PLACEBO — Sitagliptin placebo 100 mg tablet daily + Pioglitazone placebo 15 mg capsule daily
  Other Names: Januvia (sitagliptin) PLACEBO; Pioglitazone (Actos) PLACEBO
  Arms: PLACEBO

SUMMARY:
To determine whether treatment with the diabetes medication, Januvia (sitagliptin), with or without another diabetes medicine, Actos (pioglitazone), will improve insulin secretion and insulin response individuals with Impaired Glucose Tolerance (IGT), a form of prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Impaired glucose tolerance (IGT) by oral glucose tolerance test

Exclusion Criteria:

* History of diabetes mellitus
* History of congestive heart failure
* History of coronary artery disease or other macrovascular disease (stroke, peripheral vascular disease)
* History of liver disease (ALT or AST >2.5 times the upper limit of normals)
* History of renal disease (serum creatinine >1.5 mg/dl)
* History of severe osteoporosis (frequent fractures, failure on osteoporosis treatment)
* Current treatment with glucocorticoids
* History of immune disorder, including HIV
* Women of child-bearing age who are pregnant, desire to become pregnant, are breastfeeding, or who refuse to take the recommended birth control measures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Rhee, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

REFERENCES:
- [Derived] Ipsen EO, Madsen KS, Chi Y, Pedersen-Bjergaard U, Richter B, Metzendorf MI, Hemmingsen B. Pioglitazone for prevention or delay of type 2 diabetes mellitus and its associated complications in people at risk for the development of type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD013516. doi: 10.1002/14651858.CD013516.pub2. PMID 33210751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 3 control (normal glucose tolerance) subjects were enrolled to obtain results in normal subjects for the hyperglycemic clamp (without GLP-1 or arginine). No samples were run, and, therefore, there are no data for the control subjects.
  No subjects with impaired glucose tolerance (IGT) were recruited or enrolled in the study.
Period: Overall Study
Arm/Group | Sitagliptin + Pioglitazone PLACEBO | Sitagliptin + Pioglitazone | PLACEBO
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin + Pioglitazone PLACEBO | Sitagliptin + Pioglitazone | PLACEBO | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: participants]
Sex: Female, Male [Count of Participants; unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Insulin Secretion
Description: Not measured as study was prematurely terminated due to unanticipated delays.
Time Frame: baseline, 6 months, 9 months (after a 3 month washout)
Arm/Group | Sitagliptin + Pioglitazone PLACEBO | Sitagliptin + Pioglitazone | PLACEBO
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Sitagliptin + Pioglitazone PLACEBO | Sitagliptin + Pioglitazone | PLACEBO
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No